CLINICAL TRIAL: NCT05955716
Title: The Effect of Relaxation Exercise Applied With Virtual Reality Glasses on Episiotomy-induced Perineal Pain Score and Fear: A Single-Blind Randomized Controlled Study
Brief Title: Relaxation Exercise With Virtual Reality Glasses and Episiotomy-induces Perineal Pain and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem Çiçek (Other)
Collaborators: Izmir Bakircay University (Other)
Responsible Party: Sponsor-Investigator, Özlem Çiçek, Health Science Faculty Department of Nursing, Izmir Bakircay University
Organization: Izmir Bakircay University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-660
Record Dates: First submitted 2023-05-23; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Episiotomy Wound
Keywords: virtual reality glasses; episiotomy; pain; fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Experimental): During the episiotomy incision and repair, women in this group watched a relaxation video with virtual reality glasses.
  Interventions: Device: Virtual reality glasses
- Control Group (No Intervention): Women in this group received routine care in the hospital.

INTERVENTIONS:
Device: Virtual reality glasses — Virtual reality glasses are a device suitable for every mobile phone. It is used to watch the 360 degree video selected from the Youtube program.
  Arms: Virtual reality glasses

SUMMARY:
The aim of this clinical study is to compare the pain and fear scores of women who gave birth for the first time and who did and did not do relaxation exercises with virtual reality glasses during episiotomy incision and episiotomy repair.

This research seeks answers to the following questions:

Question 1: Does doing relaxation exercise with virtual reality glasses reduce the pain score experienced during episiotomy incision? Question 2: Does relaxation exercise with virtual reality glasses reduce the pain score experienced during episiotomy repair? Question 3: Does doing relaxation exercise with virtual reality glasses reduce the fear score experienced during episiotomy incision? Question 4: Does doing relaxation exercise with virtual reality glasses reduce the fear score experienced during episiotomy repair? A group of participants will be given a relaxation exercise with virtual reality glasses during the episiotomy incision and episiotomy repair. Women in the comparison group will not undergo any intervention during episiotomy incision and repair.

DETAILED DESCRIPTION:
This research is a single-blind, randomized controlled experimental study with pre-post and control groups. The population of the study consisted of pregnant women who applied to the Delivery Room in İzmir Bakırçay University Çiğli Training and Research Hospital Travay Birth Postpartum Service. The data pool could not be created because the sample was composed of women who applied for childbirth. In this randomized controlled trial, block randomization was applied. Because when simple randomization is applied, there may be a large difference between the numbers of subjects in the two groups when the study is completed. As the difference between the number of pregnant women in the virtual reality glasses and control groups grows, the reliability of the statistical analysis will decrease. Simple randomization is not recommended in cases where the sample size is less than 200. Although it was planned to take 38 experimental and 38 control group samples that met the inclusion criteria, the block randomization was carried out on 100 people, taking into account the exclusion criteria from the sample.

The randomization of the sample was made using the "random number generation program (Research Randomizer)". Intervention and control groups were formed by performing the randomization process by an impartial researcher who was not involved in the research. While it was known by the researchers in which group the pregnant women were, unilateral blindness was provided by not informing the pregnant women about the groups they were in. Since it is recommended in the literature that each step of randomized controlled trials should be performed according to the Consolidated Standards of Reporting Trials (CONSORT), this study was also conducted according to CONSORT. The type 1 error level of the study was determined as 5% (p=o.o5), the type II error level was 0.20 (80% power) and the effect size was 0.3 (moderate). Data were collected between December 2022 and May 2023. Data collection takes an average of 15 minutes.

Virtual Reality Glasses Group:

Pregnant women in the virtual reality glasses group who agreed to participate in the study and watch a relaxation video with virtual reality glasses were expected to answer the questions in the socio-demographic and obstetric information form during the latent phase of labor. Afterwards, they were asked about how many points of pain and fear they would experience on the VAS during the episiotomy incision and repair, on a scale of 0-10. After this form was answered, a relaxation video was watched with virtual reality glasses during the episiotomy incision and repair. After these procedures, as soon as the episiotomy incision and episiotomy repair were completed, virtual reality glasses were removed and the score of pain and fear they experienced was asked. They were asked to rate the pain and fear they experienced, giving a score between 0-10.

Control Group:

Pregnant women who agreed to participate in the study and who would be in the control group were expected to answer the questions in the socio-demographic and obstetric information form during the latent phase of labor. Afterwards, they were asked to score an estimated 0-10 score for pain and fear levels with VAS during episiotomy incision and repair. After this form was answered, no intervention was made during the episiotomy incision and repair, except routine practice. After these procedures, as soon as the episiotomy incision and episiotomy repair were completed, they were asked about the score of pain and fear they experienced. They were asked to rate the pain and fear they experienced, giving a score between 0-10.

Hypotheses:

1. H0-Relaxation exercise performed with virtual reality glasses does not affect the perineal pain score experienced while performing the episiotomy incision.

   H1- Relaxation exercise performed with virtual reality glasses reduces the perineal pain score experienced while performing the episiotomy incision.
2. H0-Relaxation exercise performed with virtual reality glasses does not affect the perineal pain score experienced during episiotomy suturing.

   H1- Relaxation exercise with virtual reality glasses reduces the perineal pain score experienced during episiotomy suturing.
3. H0-Relaxation exercise performed with virtual reality glasses does not affect the fear score experienced while performing the episiotomy incision.

   H1- Relaxation exercise performed with virtual reality glasses reduces the fear score experienced while applying the episiotomy incision.
4. H0- Relaxation exercise performed with virtual reality glasses does not affect the fear score experienced during episiotomy suturing.

H1- Relaxation exercise with virtual reality glasses reduces the fear score experienced during episiotomy suturing.

Data collection tool(s):

* Socio-demographic and Obstetric Information Form This form; age, education level, income level, marital status, body mass index, employment status, occupation, social security, place of residence, cohabitant, obstetric characteristics (pregnancy, birth, abortion, number of curettage), smoking and alcohol use, hospitalization In the application, there are questions about cervical dilatation and effacement level, previous delivery method, episiotomy application status. This form was applied to the women who will be included in the experimental and control groups during the latent phase of labor.
* Visual Analog Scale Pain Form The Visual Analog Scale is a scale developed by Price et al. in 1983 and is also used in the evaluation of episiotomy pain. VAS is 10 cm long. A minimum of 0 and a maximum of 10 points can be obtained from this scale. A score of zero indicates no pain, and a score of 10 indicates the pain felt at the highest level. The higher the score, the higher the level of pain.
* Visual Analog Scale Fear Form (VAS-FF) The visual analog scale is a valid and reliable measurement tool to measure other subjective emotions such as mood, in addition to pain. Fear of having an episiotomy is one of these mood changes. VAS is 10 cm long. A minimum of 0 and a maximum of 10 points can be obtained from this scale. She was asked to rate the score of fear experienced during episiotomy incision and repair between 0 and 10 points. A score of 0 indicates no fear, and a score of 10 indicates the highest level of fear. The higher the score, the higher the level of fear experienced.

Statistical method(s) to be used:

Data analysis will be done with SPSS 26 package program. In the evaluation of data; mean, standard deviation and percentage values will be calculated. In order to evaluate the homogeneity of the data according to the groups, the Skewness-Curtosis values will be examined and the tests to be used in the analysis will be decided. A probability value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria for the study:

* Turkish literacy
* Being 18 years or older
* First vaginal delivery
* Unattended vaginal delivery
* Not having a chronic disease
* Not having any complications during pregnancy
* Not using anesthetic drugs during labor
* Agreeing to practice relaxation with virtual reality glasses during the episiotomy incision and suture

Exclusion criteria from the study:

* Inability to read and write Turkish
* Incomplete answers to survey and scale questions
* Anesthesia at any stage of birth
* Deciding to have a cesarean delivery from vaginal delivery
* Opting out of participating in the research at any time of the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — • Turkish literacy
Enrollment: 76 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Score of pain experienced during episiotomy incision | Immediately after episiotomy incision
  She evaluated the pain experienced during the episiotomy incision with the help of a visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in the scores indicates an increase in the level of pain.
Score of pain experienced during episiotomy repair | Immediately after episiotomy repair
  She evaluated the pain experienced during the episiotomy repair with the help of visual analog scale. A minimum score of 0 and a maximum score of 10 are taken from this scale, and an increase in scores indicates an increase in the level of pain.
Score of fear experienced during episiotomy incision | Immediately after episiotomy incision
  She evaluated the fear experienced during the episiotomy incision with the help of visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in score indicates an increase in the level of fear.
Score of fear experienced during episiotomy repair | Immediately after episiotomy repair
  She evaluated the fear experienced during the episiotomy repair with the help of visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in score indicates an increase in the level of fear.

SECONDARY OUTCOMES:
Estimated score of pain experienced during episiotomy incision | Latent phase of birth
  She was asked to estimate how many points of pain he would have experienced during the episiotomy incision. She was asked to answer this question with the help of visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in the score indicates that she predicts that the pain she will experience will also be high.
Estimated score of pain experienced during episiotomy repair | Latent phase of birth
  She was asked to estimate how many points of pain he would have experienced during the episiotomy repair. She was asked to answer this question with the help of visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in the score indicates that she predicts that the pain she will experience will also be high.
Estimated score of fear experienced during episiotomy incision | Latent phase of birth
  She was asked to estimate how many points of fear she would have experienced during the episiotomy incision. She was asked to answer this question with the help of visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in the score indicates that she predicts that the fear she will experience will also be high.
Estimated score of fear experienced during episiotomy repair | Latent phase of birth
  She was asked to estimate how many points of fear she would have experienced during the episiotomy repair. She was asked to answer this question with the help of visual analog scale. A minimum of 0 and a maximum of 10 points are taken from this scale, and an increase in the score indicates that she predicts that the fear she will experience will also be high.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çiçek, PhD, Principal Investigator — Izmir Bakırçay University; Gamze Durmazoğlu, PhD, Study Chair — Izmir Ataturk Training and Research Hospital; Dilek Mamik Aktay, Msc, Study Chair — Izmir Bakırçay University Training and Research Hospital
Locations (1):
- Özlem Çiçek, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] JahaniShoorab N, Ebrahimzadeh Zagami S, Nahvi A, Mazluom SR, Golmakani N, Talebi M, Pabarja F. The Effect of Virtual Reality on Pain in Primiparity Women during Episiotomy Repair: A Randomize Clinical Trial. Iran J Med Sci. 2015 May;40(3):219-24. PMID 25999621
- [Result] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747
- [Result] Czech O, Wrzeciono A, Rutkowska A, Guzik A, Kiper P, Rutkowski S. Virtual Reality Interventions for Needle-Related Procedural Pain, Fear and Anxiety-A Systematic Review and Meta-Analysis. J Clin Med. 2021 Jul 23;10(15):3248. doi: 10.3390/jcm10153248. PMID 34362032
- [Result] Priddis H, Dahlen HG, Schmied V, Sneddon A, Kettle C, Brown C, Thornton C. Risk of recurrence, subsequent mode of birth and morbidity for women who experienced severe perineal trauma in a first birth in New South Wales between 2000-2008: a population based data linkage study. BMC Pregnancy Childbirth. 2013 Apr 8;13:89. doi: 10.1186/1471-2393-13-89. PMID 23565655
- [Result] ACOG Practice Bulletin No. 154: Operative Vaginal Delivery. Obstet Gynecol. 2015 Nov;126(5):e56-e65. doi: 10.1097/AOG.0000000000001147. No abstract available. PMID 26488523
- [Result] Kartal B, Kizilirmak A, Calpbinici P, Demir G. Retrospective analysis of episiotomy prevalence. J Turk Ger Gynecol Assoc. 2017 Dec 15;18(4):190-194. doi: 10.4274/jtgga.2016.0238. PMID 29278232
- [Result] Jiang H, Qian X, Carroli G, Garner P. Selective versus routine use of episiotomy for vaginal birth. Cochrane Database Syst Rev. 2017 Feb 8;2(2):CD000081. doi: 10.1002/14651858.CD000081.pub3. PMID 28176333
- [Result] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Result] Solt Kirca A, Korkut Oksuz S, Murat N. The effect of cold application on episiotomy pain: A systematic review and meta-analysis. J Clin Nurs. 2022 Mar;31(5-6):559-568. doi: 10.1111/jocn.15912. Epub 2021 Jun 13. PMID 34121251
- [Result] Zibanejad S, Miraj S, Rafieian Kopaei M. Healing effect of Quercus persica and Lawsonia inermis ointment on episiotomy wounds in primiparous women. J Res Med Sci. 2020 Feb 20;25:11. doi: 10.4103/jrms.JRMS_251_18. eCollection 2020. PMID 32174983